CLINICAL TRIAL: NCT03802617
Title: A Phase II Clinical Study of MR13A9 in Hemodialysis Patients With Pruritus.
Brief Title: A Clinical Study of MR13A9 in Hemodialysis Patients With Pruritus.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Collaborators: Maruishi Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MR13A9-4
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2021-02

CONDITIONS: Uremic Pruritus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MR13A9 low dose (Experimental)
  Interventions: Drug: MR13A9
- MR13A9 medium dose (Experimental)
  Interventions: Drug: MR13A9
- MR13A9 high dose (Experimental)
  Interventions: Drug: MR13A9
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MR13A9 — Intravenous administration
  Arms: MR13A9 high dose; MR13A9 low dose; MR13A9 medium dose
Drug: Placebo — Intravenous administration
  Arms: Placebo

SUMMARY:
Double-blind, Placebo-controlled study to evaluate the dose-response relationship of safety, efficacy and pharmacokinetics of MA13A9 in hemodialysis patients with pruritus.

ELIGIBILITY:
Inclusion Criteria:

* Japanese with male or female aged ≥ 20
* Patient with Chronic Kidney Disease (CKD) has been on hemodialysis 3 times per week
* Patient receiving treatment for itch
* Patient has a baseline NRS score > 4

Exclusion Criteria:

* Patient has pruritus cause other than CKD or its complications
* Patients has hepatic cirrhosis
* Patient has a known history of allergic reaction to opiates

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2019-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Koshihara, Study Director — Clinical Development Div.
Locations (1):
- Research Site, Multiple Locations, Japan

REFERENCES:
- [Derived] Narita I, Tsubakihara Y, Uchiyama T, Okamura S, Oya N, Takahashi N, Gejyo F; MR13A9-4 Trial Investigators. Efficacy and Safety of Difelikefalin in Japanese Patients With Moderate to Severe Pruritus Receiving Hemodialysis: A Randomized Clinical Trial. JAMA Netw Open. 2022 May 2;5(5):e2210339. doi: 10.1001/jamanetworkopen.2022.10339. PMID 35511180

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 311 participants who had been screened, 247 subjects were enrolled in this study and were randomly assigned to each study drugs. 225 subjects completed the study and 22 subjects discontinued the study.
Groups:
- 0.25 μg/kg Group: The study drug was injected into the venous line of the dialysis circuit at the end of each dialysis session for 8 weeks (3 times weekly, 24 times in total). The injected volume of the study drug was determined based on the subject's dry weight on the day of dosing as below.
  * < 45.0 kg: 8.75 μg
  * >= 45.0 kg, < 65.0 kg: 12.50 μg
  * >= 65.0 kg, < 85.0 kg: 17.50 μg
  * >= 85.0 kg: 21.25 μg
- 0.5 μg/kg Group: The study drug was injected into the venous line of the dialysis circuit at the end of each dialysis session for 8 weeks (3 times weekly, 24 times in total). The injected volume of the study drug was determined based on the subject's dry weight on the day of dosing as below.
  * < 45.0 kg: 17.5 μg
  * >= 45.0 kg, < 65.0 kg: 25.0 μg
  * >= 65.0 kg, < 85.0 kg: 35.0 μg
  * >= 85.0 kg: 42.5 μg
- 1.0 μg/kg Group: The study drug was injected into the venous line of the dialysis circuit at the end of each dialysis session for 8 weeks (3 times weekly, 24 times in total). The injected volume of the study drug was determined based on the subject's dry weight on the day of dosing as below.
  * < 45.0 kg: 35.0 μg
  * >= 45.0 kg, < 65.0 kg: 50.0 μg
  * >= 65.0 kg, < 85.0 kg: 70.0 μg
  * >= 85.0 kg: 85.0 μg
- Placebo Group: The study drug was injected into the venous line of the dialysis circuit at the end of each dialysis session for 8 weeks (3 times weekly, 24 times in total).
Period: Overall Study
Arm/Group | 0.25 μg/kg Group | 0.5 μg/kg Group | 1.0 μg/kg Group | Placebo Group
Started | 61 | 61 | 62 | 63
Completed | 59 | 53 | 54 | 59
Not Completed | 2 | 8 | 8 | 4
Not completed — Adverse Event | 0 | 4 | 5 | 1
Not completed — Lack of Efficacy | 0 | 1 | 0 | 2
Not completed — Protocol Violation | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0
Not completed — Four consecutive missed doses of the study drug | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: One subject of 1.0 μg/kg group was excluded from FAS due to deviation from one of the inclusion criteria. So, there is a discrepancy between the number of subjects in "Participant flow" and in "Overall Number of Baseline Participants".
Groups:
- 1.0 μg/kg Group: The study drug will be injected into the venous line of the dialysis circuit at the end of each dialysis session for 8 weeks (3 times weekly, 24 times in total). The injected volume of the study drug was determined based on the subject's dry weight on the day of dosing as below.
  * < 45.0 kg: 35.0 μg
  * >= 45.0 kg, < 65.0 kg: 50.0 μg
  * >= 65.0 kg, < 85.0 kg: 70.0 μg
  * >= 85.0 kg: 85.0 μg
- Total: Total of all reporting groups
Arm/Group | 0.25 μg/kg Group | 0.5 μg/kg Group | 1.0 μg/kg Group | Placebo Group | Total
Number analyzed (Participants) | 61 | 61 | 61 | 63 | 246
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 25 | 29 | 30 | 107
  >=65 years | 38 | 36 | 32 | 33 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (11.2) | 65.6 (11.4) | 64.4 (11.7) | 64.1 (12.7) | 64.5 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 16 | 14 | 20 | 61
  Male | 50 | 45 | 47 | 43 | 185
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 61 | 61 | 61 | 63 | 246
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 61 | 61 | 61 | 63 | 246
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 61 | 61 | 61 | 63 | 246
Dry weight at the start of Sceening [Mean (Standard Deviation); unit: kg] | 61.25 (13.86) | 59.98 (11.22) | 62.85 (13.39) | 60.63 (12.71) | 61.17 (12.80)
Hemodialysis History [Mean (Standard Deviation); unit: years] | 7.0 (6.5) | 6.7 (7.2) | 7.7 (6.5) | 6.8 (6.1) | 7.1 (6.5)
Disease duration of Itch [Mean (Standard Deviation); unit: years] | 3.7 (3.5) | 4.5 (4.4) | 4.8 (4.9) | 4.3 (4.4) | 4.3 (4.3)
Average NRS Score [Mean (Standard Deviation); unit: points] — Looking back on the period between the time of awakening on the previous day of assessment and the time of awakening on the day of assessment (including sleeping hours) once daily, subjects will assess the NRS score for the most severe itching by themselves. The most severe itching within the day will be assessed in integer on a scale ranging from 0 to 10, where 0 represents no itching and 10 represents worst itching imaginable.
  points | 6.35 (1.24) | 6.83 (1.40) | 6.47 (1.29) | 6.53 (1.31) | 6.55 (1.31)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Mean NRS Score at Week 8 of the Treatment Period
Description: The primary analysis was performed using an MMRM with change from baseline in the mean NRS score at each time point as an objective variable; treatment group, time point, and treatment group-by-time point interaction as fixed effects; baseline mean NRS score and dynamic allocation factors, presence of prior treatment with nalfurafine hydrochloride, and presence of specific signs or symptoms to be confirmed in the screening period, as covariates; and subject as a random effect.
  Looking back on the period between the time of awakening on the previous day of assessment and the time of awakening on the day of assessment (including sleeping hours) once daily, subjects will assess the NRS score for the most severe itching by themselves. The most severe itching within the day will be assessed in integer on a scale ranging from 0 to 10, where 0 represents no itching and 10 represents worst itching imaginable.
Time Frame: 8 weeks
Population: One subject of 1.0 μg/kg group was excluded from FAS due to deviation from one of the inclusion criteria. So, there is a discrepancy between the number of subjects in "Participant flow" and in "Overall Number of Participants Analyzed".
Measure: Mean (Standard Error); unit: points
Arm/Group | 0.25 μg/kg Group | 0.5 μg/kg Group | 1.0 μg/kg Group | Placebo Group
Number analyzed (Participants) | 61 | 61 | 61 | 63
points | -2.97 (0.29) | -3.65 (0.30) | -3.64 (0.30) | -2.86 (0.29)
Statistical Analysis 1: Comparison: 0.25 μg/kg Group vs Placebo Group; Test type: Other; p = 0.770, MMRM; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.85 to 0.63], Standard Error of Mean 0.38
Statistical Analysis 2: Comparison: 0.5 μg/kg Group vs Placebo Group; Test type: Other; p = 0.038, MMRM; Mean Difference (Final Values) = -0.80, 95% CI 2-sided [-1.55 to -0.04], Standard Error of Mean 0.38
Statistical Analysis 3: Comparison: 1.0 μg/kg Group vs Placebo Group; Test type: Other; p = 0.041, MMRM; Mean Difference (Final Values) = -0.78, 95% CI 2-sided [-1.54 to -0.03], Standard Error of Mean 0.38

ADVERSE EVENTS:
Time Frame: Up to 8 weeks
Arm/Group | 0.25 μg/kg Group | 0.5 μg/kg Group | 1.0 μg/kg Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/61 | 0/62 | 0/63
Serious Adverse Events (participants affected / at risk) | 3/61 | 8/61 | 5/62 | 2/63
Other Adverse Events (participants affected / at risk) | 30/61 | 35/61 | 40/62 | 24/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.25 μg/kg Group (N=61) | 0.5 μg/kg Group (N=61) | 1.0 μg/kg Group (N=62) | Placebo Group (N=63)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitreous opacities (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heat illness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shunt malfunction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shunt occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shunt stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.25 μg/kg Group (N=61) | 0.5 μg/kg Group (N=61) | 1.0 μg/kg Group (N=62) | Placebo Group (N=63)
Constipation (Gastrointestinal disorders) | 5 (5) | 3 (3) | 7 (7) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (5) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (5) | 3 (3)
Malaise (General disorders) | 2 (2) | 2 (2) | 4 (5) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 8 (8) | 6 (8) | 3 (3) | 7 (8)
Procedural hypotension (Injury, poisoning and procedural complications) | 4 (7) | 3 (3) | 2 (3) | 3 (4)
Blood pressure decreased (Investigations) | 0 (0) | 4 (4) | 3 (3) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (7) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 3 (3) | 5 (5) | 3 (4)
Somnolence (Nervous system disorders) | 2 (2) | 3 (3) | 6 (6) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/17/NCT03802617/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT03802617/SAP_001.pdf